CLINICAL TRIAL: NCT06095596
Title: Efficacy and Safety Analysis of Sequential Treatment of Moderate to Severe Ulcerative Colitis With Vedolizumab and Upadacitinib: A Multicenter Prospective Randomized Controlled Clinical Study
Brief Title: Efficacy and Safety of Vedolizumab Combined With Upadacitinib in Patients With Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jiayin Yao, Principal investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZSLYEC-469
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis (UC)
MeSH Terms: conditions — Colitis, Ulcerative | interventions — upadacitinib; vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination treatment group (Experimental): A combination treatment of vedolizumab and upadacitinib for 8 weeks in the induction therapy, then followed by a single treatment of vedolizumab in the maintenance therapy
  Interventions: Drug: Upadacitinib; Drug: Vedolizumab
- Single treatment group (Placebo Comparator): single treatment of vedolizumab both in the induction and maintenance therapy
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Upadacitinib — Oral upadacitinib 45mg/d for 8 weeks in the induction therapy.
  Other Names: Upadacitinib treatment
  Arms: Combination treatment group
Drug: Vedolizumab — Vedolizumab 300mg intravenously on weeks 1, 2, 6, and then on every 8-week interval.
  Other Names: Vedolizumab treatment

SUMMARY:
It's of great importance to effectively induce and maintain disease remission in patients with moderate to severe ulcerative colitis (UC). Vedolizumab (VDZ) is known for its high safety profile and confirmed therapeutic efficacy in UC treatment. However, according to the experience in clinical practice, the effect onset speed of vedolizumab is relatively slow. Upadacitinib (UPA), however, works quickly, which complements the defect of slow onset of VDZ induction. However, the safety of UPA used in situations such as infection and tumors is inferior to that of VDZ, and long-term use requires testing for the risk of adverse events such as deep vein thrombosis. Therefore, if the advantages of long-term maintenance therapy safety of VDZ and rapid induced remission of UPA are fully utilized, the combination of VDZ and UPA induction for 8 weeks, followed by the use of single drug VDZ in maintenance therapy, can maximize the clinical benefits of UC patients. Due to the lack of high-level clinical research data at home and abroad, we plan to conduct a multicenter prospective randomized controlled clinical study to provide the evidence-based basis for the efficacy analysis of the sequential treatment of moderate to severe UC patients with VDZ and UPA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed UC for at least 3 months, including endoscopic evidence supporting UC and histopathological evidence supporting UC diagnosis
* Suffering from moderate to severe UC, defined as modified Mayo score ≥ 4 and endoscopic subscale (ESS) ≥ 2
* Indications for VDZ or UPA application

Exclusion Criteria:

* Patients who are unable to take oral UPA and receive regular intravenous VDZ infusion therapy
* Evidence of toxic megacolon was found during screening
* Previously underwent extensive colectomy, subtotal resection, or total colectomy, ileostomy, or colostomy due to UC
* Subjects who require surgery due to UC or plan to undergo elective surgery during the study period
* There is evidence indicating that the subjects suffer from severe, progressive, or uncontrolled kidney, liver, blood, endocrine, respiratory, mental, or neurological diseases
* Evidence of active hepatitis B or C infection during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
8th-week endoscopic remission rate | 8th-week
  endoscopic subscale (ESS) =0, which defined as endoscopic remission

SECONDARY OUTCOMES:
Clinical remission rate at the 8th week | 8th-week
  Clinical remission is defined as a total Mayo score ≤2, with no individual subscore >1 and a rectal bleeding subscore of 0.
clincial response rate at 8th-week | 8th-week
  Clinical response is defined as a decrease in total Mayo score by ≥3 points and ≥30% from baseline, with a decrease in rectal bleeding subscore by ≥1 point or an absolute rectal bleeding subscore of 0 or 1.
Endoscopic response rate at 8th-week | 8th-week
  Endoscopic response is defined as a decrease in the Mayo endoscopic subscore by ≥1 point from baseline
normalization rate of CRP at the 8th week | 8th-week
  normalization rate of C reactive protein (CRP)
life quality score at the 8th week | 8th-week
  Inflammatory bowel disease questionnaire (IBDQ), the total score is 32-224, with higher scores indicating better quality of life for patients.
Clinical remission rate at the 54th-week | 54th-week
  clincial remisson is defined as a total Mayo score ≤2, with no individual subscore >1 and a rectal bleeding subscore of 0.
Clinical response rate at 54th week | 54th week
  Clinical response is defined as a decrease in total Mayo score by ≥3 points and ≥30% from baseline, with a decrease in rectal bleeding subscore by ≥1 point or an absolute rectal bleeding subscore of 0 or 1.
endoscopic remission rate at 54th-week | 54th-week
  endoscopic subscale (ESS) =0, which defined as endoscopic remission
Endoscopic response rate at 54th-week | 54th-week
  Endoscopic response is defined as a decrease in the Mayo endoscopic subscore by ≥1 point from baseline
normalization rate of CRP at the 54th week | 54th-week
  normalization rate of CRP
life quality score at the 54th week | 54th-week
  Inflammatory bowel disease questionnaire (IBDQ), the total score is 32-224, with higher scores indicating better quality of life for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No